CLINICAL TRIAL: NCT06400433
Title: Comparison of the Efficacy of Ultrasound-Guided Median Nerve Hydrodissection With Dexamethasone and Dextrose at Different Volumes in Patients With Carpal Tunnel Syndrome: A Prospective, Randomized, Double Blind Study
Brief Title: Comparing Efficacies of Median Nerve Hydrodissection With Dexamethasone and Dextrose in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sevgi Selin Kurtoglu, Residency doctor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IstanbulUC-SKurtoglu-01
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Carpal Tunnel Syndrome; Median Nerve Entrapment; Entrapment Neuropathy
Keywords: Median nerve hydrodissection; Ultrasound guided injection
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy; Charcot-Marie-Tooth Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient, the administering physician, the physician conducting the clinical and ultrasonographic evaluation, and the physician performing the electrophysiological examination will not be informed about the injection materials assigned to the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 5 ml of %5 dextrose (Active Comparator): The physical examination, handgrip strength values, two-point discrimination, pain scoring (numeric rating scale), Q-DASH, BCTQ, CTS-6 scores, and ultrasonographically measured median nerve cross-sectional area values of the patients in this group will be evaluated and recorded by the first physician before the treatment and at the second, fourth, and twelfth weeks. The nerve conduction study will be examined by the second physician before the treatment and at the twelfth week.
  Patients in this group will be treated with ultrasound-guided median nerve hydrodissection by in-plane technique with 5 ml of %5 dextrose solution.
  Interventions: Procedure: Ultrasound-guided median nerve hydrodissection
- 10 ml of %5 dextrose (Active Comparator): The physical examination, handgrip strength values, two-point discrimination, pain scoring (numeric rating scale), Q-DASH, BCTQ, CTS-6 scores, and ultrasonographically measured median nerve cross-sectional area values of the patients in this group will be evaluated and recorded by the first physician before the treatment and at the second, fourth, and twelfth weeks. The nerve conduction study will be examined by the second physician before the treatment and at the twelfth week.
  Patients in this group will be treated with ultrasound-guided median nerve hydrodissection by in-plane technique with 10 ml of %5 dextrose solution.
  Interventions: Procedure: Ultrasound-guided median nerve hydrodissection
- 2 ml of 8 mg dexamethasone + 3 ml normal saline (Active Comparator): The physical examination, handgrip strength values, two-point discrimination, pain scoring (numeric rating scale), Q-DASH, BCTQ, CTS-6 scores, and ultrasonographically measured median nerve cross-sectional area values of the patients in this group will be evaluated and recorded by the first physician before the treatment and at the second, fourth, and twelfth weeks. The nerve conduction study will be examined by the second physician before the treatment and at the twelfth week.
  Patients in this group will be treated with ultrasound-guided median nerve hydrodissection by in-plane technique with 2 ml of 8 mg dexamethasone + 3 ml %0,9 NaCl solution (normal saline).
  Interventions: Procedure: Ultrasound-guided median nerve hydrodissection
- 2 ml of 8 mg dexamethasone + 8 ml normal saline (Active Comparator): The physical examination, handgrip strength values, two-point discrimination, pain scoring (numeric rating scale), Q-DASH, BCTQ, CTS-6 scores, and ultrasonographically measured median nerve cross-sectional area values of the patients in this group will be evaluated and recorded by the first physician before the treatment and at the second, fourth, and twelfth weeks. The nerve conduction study will be examined by the second physician before the treatment and at the twelfth week.
  Patients in this group will be treated with ultrasound-guided median nerve hydrodissection by in-plane technique with 2 ml of 8 mg dexamethasone + 8 ml %0,9 NaCl solution (normal saline).
  Interventions: Procedure: Ultrasound-guided median nerve hydrodissection

INTERVENTIONS:
Procedure: Ultrasound-guided median nerve hydrodissection — Injected wrist will be supinated and slightly dorsiflexed. The transducer of the ultrasound will be placed transversely at the proximal carpal inlet. After sterile preparation, a 22 gauge needle will be inserted using the short-axis technique, in-plane ulnar approach. During hydrodissection, separation of either between the median nerve and flexor retinaculum or between the median nerve and the underlying flexor tendons will be visually confirmed.

SUMMARY:
The aim of this study is to compare the efficacy of ultrasonography-guided hydrodissection technique with 5% dextrose and dexamethasone injectates when applied in different volumes in the treatment of mild to moderate carpal tunnel syndrome.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common peripheral nerve entrapment neuropathy worldwide, resulting from the compression of the median nerve in the carpal tunnel, an osteofibrous canal whose roof is formed by the flexor retinaculum and whose floor is formed by the carpal bones. CTS accounts for approximately 90% of all entrapment neuropathies, and an individual's lifetime risk of diagnosis is estimated to be 10%. It is estimated that about 5% of the population suffers from CTS. It is more common in women compared to men and at least half of the cases manifests between the ages of 40 and 60.

In clinical practice, the most common complaints of patients include neuropathic symptoms along the distribution of the median nerve. These complaints, which initially occur and flare up at night and intermittently during the day, may become continuous and worsen in the later stages of the disease.

Taking an accurate history and clinical assessment is crucial for diagnosis. Evaluation of sensory abnormalities, loss of two point discrimination, and the strength of abductor pollicis brevis muscle can provide information about functional impairment. Tinel's sign and Phalen's manoeuvre are some of diagnostic tests. Some scales and questionnaires are used in diagnosis and assessment of functionality. Ultrasonography is a useful, inexpensive and easily accessible method to simultaneously observe morphological changes in the median nerve and scan the surrounding anatomy. Electrophysiological assessment is very sensitive in examining median nerve dysfunction caused by nerve damage. Nerve conduction studies are considered the gold standard method in diagnosis, determining prognosis and making treatment decisions.

The management of CTS in patients depends on the severity of the disease. In mild and moderate circumstances conservative treatments are recommended for the patients. Surgery is typically considered for patients with moderate to severe CTS or individuals who do not experience significant improvement with conservative treatments. Conservative treatments include patient education, wrist splinting, medical treatments, physical therapy, and perineural injections.

Ultrasound-guided nerve hydrodissection injection has emerged as a therapeutic approach with less complications for CTS. This method aims to achieve mechanical release from perineural adhesions by creating a perineural fluid plane.Various injectates such as normal saline, 5% dextrose, and platelet-rich plasma,viscosupplements are commonly used for hydrodissection. Many studies have been conducted with the hypothesis that the injection volume, in addition to the injection preparation, would also be important in median nerve hydrodissection, and different results have been obtained.

This study aimed to compare the clinical, ultrasonographic and electrophysiological improvement in patients by applying different volumes of dexamethasone and dextrose in median nerve hydrodissection. Patients will be evaluated before and after treatment at 2nd, 4th and 12th weeks ultrasonographically, electrophysiologically and clinically with pain scores, handgrip strength assesment, two-point discrimination values, functional and disability scales.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age or older
* Patients who are clinically diagnosed with CTS
* Patients who have mild or moderate CTS confirmed by EMG study
* Patients unresponsive to 2-weeks of nightly volar wrist splinting

Exclusion Criteria:

* Patients who are younger than 18 years of age
* Patients with severe EMG study
* Presence of thenar atrophy
* Patients diagnosed with cervical radiculopathy, myelopathy, brachial plexopathy or polyneuropathy
* Patients diagnosed with thoracic outlet syndrome
* Patients diagnosed with inflammatory rheumatic disease
* Patients diagnosed with connective tissue disease
* Patients diagnosed with neuromuscular disease
* Patients diagnosed with peripheral vascular disease
* Patients with history of malignancy
* Patients who have uncontrolled hypothyroidism, hyperthyroidism or diabetes mellitus
* Patients diagnosed with chronic renal failure
* Patients diagnosed with acromegaly
* Patients with history of surgery and/or fracture at the symptomatic upper extremity
* Patients with a history of injection into the median nerve lasting less than 6 months at the symptomatic wrist
* Patients who are pregnant
* Patients with history of chronic steroid or chronic alcohol use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical improvement measured by change in Numeric Rating Scale | Baseline, 2nd week, 4th week, 12th week
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. Scale ranges from '0' representing "no pain" to '10' representing "pain as bad as you can imagine" or "worst pain imaginable". Higher scores related to worse outcome.
Functional and clinical improvement measured by change in Quick- Disabilities of Arm, Shoulder and Hand Questionnaire (Q-DASH) Scores | Baseline, 2nd week, 4th week, 12th week
  The Q-DASH questionnaire, which is a shortened version of the DASH questionnaire, consists of 11 items to measure physical functions and symptoms of the upper extremity. In order for the Q-DASH score to be calculated, at least 10 of the 11 topics must be answered. All items are scored between 1-5. In this scoring, 1 point indicates not having any difficulty during the activity, while 5 points indicates not being able to do the activity at all. Calculating the total score as 0 (zero) indicates no disability, while the highest score of 100 indicates the highest disability.
  In our study, the investigator will use the Turkish form of the Q-DASH questionnaire, whose validity and reliability has been demonstrated.
Change in median nerve cross-sectional area values | Baseline, 2nd week, 4th week, 12th week
  The median nerve cross-sectional area value will be measured by ultrasound at the proximal inlet of the carpal tunnel at the level of the os pisiforme and os hamatum.
Functional and clinical improvement measured by change in Boston Carpal Tunnel Questionnaire (BCTQ) | Baseline, 2nd week, 4th week, 12th week
  It is a symptom and functionality assessment questionnaire for carpal tunnel syndrome developed by Levine et al. in 1993. It consists of two parts that evaluate symptom severity (Symptom Severity Scale) and functional status (Functional Status Scale). It consists of 11 questions about symptoms and 8 questions about functional status and has 5 possible answers. Each answer is scored between 1-5. The two sections are evaluated separately and the total score obtained. Minimum Symptom Severity Scale score is 11 and maximum score is 55. Minimum Functional Status Scale score is 8 and maximum score is 40. Calculating the total score as 19 (nineteen) indicates no disability, while the highest score of 95 (ninety five) indicates the highest disability.
  In our study, the investigator will use the Turkish language version of BCTQ, the validity and reliability of which has been demonstrated.
Change in median sensory nerve latency (SNL) values from the electrophysiological study | Baseline, 12th week
  Electrophysiological Study: Sensory and motor nerve conduction studies of both median and ulnar nerve
Change in median nerve distal motor latency (DML) values from the electrophysiological study | Baseline, 12th week
  Electrophysiological Study: Sensory and motor nerve conduction studies of both median and ulnar nerve
Change in median sensory nerve action potential (SNAP) values from the electrophysiological study | Baseline, 12th week
  Electrophysiological Study: Sensory and motor nerve conduction studies of both median and ulnar nerve
Change in median nerve compound muscle action potential (CMAP) values from the electrophysiological study | Baseline, 12th week
  Electrophysiological Study: Sensory and motor nerve conduction studies of both median and ulnar nerve
Change in median motor nerve conduction velocity (MNCV) values from the electrophysiological study | Baseline, 12th week
  Electrophysiological Study: Sensory and motor nerve conduction studies of both median and ulnar nerve
Change in median sensory nerve conduction velocity (SNCV) values from the electrophysiological study | Baseline, 12th week
  Electrophysiological Study: Sensory and motor nerve conduction studies of both median and ulnar nerve
Change in 6-item CTS symptoms scale scores | Baseline, 2nd week, 4th week, 12th week
  It consists of 6 items. A special score was created for each item. The score of each item is calculated by addition. Minimum score is 0 (zero), maximum score is 26 (twenty six). Patients who score 12 points or more in total are highly expected to have CTS.

SECONDARY OUTCOMES:
Change in hand grip strength values | Baseline, 2nd week, 4th week, 12th week
  Measured by Jamar hand dynomometry, scored in kilograms, higher scores indicate better outcomes
Change in two point discrimination test values | Baseline, 2nd week, 4th week, 12th week
  Measured 4-8 mm, higher than 5 mm score considered abnormal discrimination and higher scores indicates worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi S Kurtoglu, MD, Principal Investigator — Istanbul University - Cerrahpasa; Kenan Akgun, MD, Study Director — Istanbul University - Cerrahpasa; Rana Terlemez, MD, Study Chair — Istanbul University - Cerrahpasa; Jale Zare, MD, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa (IUC), Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padua L, Coraci D, Erra C, Pazzaglia C, Paolasso I, Loreti C, Caliandro P, Hobson-Webb LD. Carpal tunnel syndrome: clinical features, diagnosis, and management. Lancet Neurol. 2016 Nov;15(12):1273-1284. doi: 10.1016/S1474-4422(16)30231-9. Epub 2016 Oct 11. PMID 27751557
- [Background] Mondelli M, Giannini F, Giacchi M. Carpal tunnel syndrome incidence in a general population. Neurology. 2002 Jan 22;58(2):289-94. doi: 10.1212/wnl.58.2.289. PMID 11805259
- [Background] Atroshi I, Gummesson C, Johnsson R, Ornstein E, Ranstam J, Rosen I. Prevalence of carpal tunnel syndrome in a general population. JAMA. 1999 Jul 14;282(2):153-8. doi: 10.1001/jama.282.2.153. PMID 10411196
- [Background] Padua L, Padua R, Lo Monaco M, Aprile I, Tonali P. Multiperspective assessment of carpal tunnel syndrome: a multicenter study. Italian CTS Study Group. Neurology. 1999 Nov 10;53(8):1654-9. doi: 10.1212/wnl.53.8.1654. PMID 10563608
- [Background] Wong SM, Griffith JF, Hui AC, Lo SK, Fu M, Wong KS. Carpal tunnel syndrome: diagnostic usefulness of sonography. Radiology. 2004 Jul;232(1):93-9. doi: 10.1148/radiol.2321030071. Epub 2004 May 20. PMID 15155897
- [Background] Fowler JR, Gaughan JP, Ilyas AM. The sensitivity and specificity of ultrasound for the diagnosis of carpal tunnel syndrome: a meta-analysis. Clin Orthop Relat Res. 2011 Apr;469(4):1089-94. doi: 10.1007/s11999-010-1637-5. Epub 2010 Oct 21. PMID 20963527
- [Background] Padua L, LoMonaco M, Gregori B, Valente EM, Padua R, Tonali P. Neurophysiological classification and sensitivity in 500 carpal tunnel syndrome hands. Acta Neurol Scand. 1997 Oct;96(4):211-7. doi: 10.1111/j.1600-0404.1997.tb00271.x. PMID 9325471
- [Background] Padua L, LoMonaco M, Aulisa L, Tamburrelli F, Valente EM, Padua R, Gregori B, Tonali P. Surgical prognosis in carpal tunnel syndrome: usefulness of a preoperative neurophysiological assessment. Acta Neurol Scand. 1996 Nov;94(5):343-6. doi: 10.1111/j.1600-0404.1996.tb07077.x. PMID 8947287
- [Background] Jablecki CK, Andary MT, So YT, Wilkins DE, Williams FH. Literature review of the usefulness of nerve conduction studies and electromyography for the evaluation of patients with carpal tunnel syndrome. AAEM Quality Assurance Committee. Muscle Nerve. 1993 Dec;16(12):1392-414. doi: 10.1002/mus.880161220. PMID 8232399
- [Background] Ostergaard PJ, Meyer MA, Earp BE. Non-operative Treatment of Carpal Tunnel Syndrome. Curr Rev Musculoskelet Med. 2020 Apr;13(2):141-147. doi: 10.1007/s12178-020-09616-0. PMID 32124335
- [Background] Malone DG, Clark TB, Wei N. Ultrasound-guided percutaneous injection, hydrodissection, and fenestration for carpal tunnel syndrome: description of a new technique. J Appl Res. (2010) 10:117.
- [Background] Evers S, Thoreson AR, Smith J, Zhao C, Geske JR, Amadio PC. Ultrasound-guided hydrodissection decreases gliding resistance of the median nerve within the carpal tunnel. Muscle Nerve. 2018 Jan;57(1):25-32. doi: 10.1002/mus.25723. Epub 2017 Jul 6. PMID 28622409
- [Background] Lin MT, Liao CL, Hsiao MY, Hsueh HW, Chao CC, Wu CH. Volume Matters in Ultrasound-Guided Perineural Dextrose Injection for Carpal Tunnel Syndrome: A Randomized, Double-Blinded, Three-Arm Trial. Front Pharmacol. 2020 Dec 17;11:625830. doi: 10.3389/fphar.2020.625830. eCollection 2020. PMID 33391002
- [Background] Buntragulpoontawee M, Chang KV, Vitoonpong T, Pornjaksawan S, Kitisak K, Saokaew S, Kanchanasurakit S. The Effectiveness and Safety of Commonly Used Injectates for Ultrasound-Guided Hydrodissection Treatment of Peripheral Nerve Entrapment Syndromes: A Systematic Review. Front Pharmacol. 2021 Mar 5;11:621150. doi: 10.3389/fphar.2020.621150. eCollection 2020. PMID 33746745